CLINICAL TRIAL: NCT03261622
Title: Sacral Nerve Stimulation for Faecal Incontinence - Placebo or Clinical Effective: A Randomized Blinded Study
Brief Title: Sacral Nerve Stimulation for Faecal Incontinence - Placebo or Clinical Effective
Acronym: SNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Tromso (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Jakobsen, Principal Investigator (M.D. Ph.D.), University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 005
Record Dates: First submitted 2017-06-23; First posted 2017-08-25 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Faecal Incontinence; Fecal Incontinence
Keywords: Sacral Nerve Stimulation; Sacral Nerve Modulation
MeSH Terms: conditions — Encopresis; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either control group (Stimulation amplitude at 90% of sensory threshold) or intervention arm (different stimulation amplitude - 0.05 V, 50 and 90% of sensory threshold)
Who Masked: Participant, Investigator
Masking Description: Alle patients are stimulated sub-sensory in (3x4 weeks) and will be blinded. The investigators will not participate in the randomization, and setting of the stimulation amplitude.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Stimulation amplitude at 90% of sensory threshold during period 1 to 3. (each period 4 weeks)
  Interventions: Device: Sacral nerve stimulation at different stimulation amplitudes
- Intervention arm (Sham Comparator): Alternation of stimulation amplitude
  1. Period - Stimulation amplitude 0.05 Volts (lowest possible)
  2. Period - Stimulation amplitude - 50% of sensory threshold.
  3. Period - Stimulation amplitude - 90% of sensory threshold.
  Interventions: Device: Sacral nerve stimulation at different stimulation amplitudes

INTERVENTIONS:
Device: Sacral nerve stimulation at different stimulation amplitudes — Exploring the effect of different stimulation amplitude in a randomized study

SUMMARY:
Sacral nerve stimulation (SNS) has over the last 20 years been recognised as an efficient treatment option for faecal incontinence (FI).

In a selected patient group we have evidence that 90% of patients will have a successful test period (≥50% reduction in incontinence episodes). If preoperative there is motor response on at least 3 out of 4 poles on the lead, at a threshold ≤1.5 mAMP.

Hypotheses In a selected patient group suffering from faecal incontinence a one-stage permanent implant will be possible. The functional results will be improved as more time can be spent finding the optimal pacemaker settings as the risk of infection is reduced compared to the stage implant. One-Stage implantation gives the opportunity to test the amount of placebo effect with SNS.

During the first 3 months postoperative patients will be randomized to either stimulation amplitude set at 90% of sensory threshold (control group) or 3 periods of stimulation at 0.05v (placebo), 50% and 90% of sensory threshold. Patients are randomized in a 1 to 2 pattern. After the initial 3 months the stimulation amplitude is increased to sensory threshold. After six months the project ends and the number of patients achieving the 50% improvement in incontinence episodes are evaluated.

DETAILED DESCRIPTION:
Sacral nerve stimulation (SNS) has over the last 20 years been recognised as an efficient treatment option for faecal incontinence (FI). The therapy is recommended by the International Continence Society (ICS) if conservative treatments such as; regulation of diet and fibre supplements, medication, biofeedback therapy, glycerol suppositories, mini enema or transanal irrigation have been insufficient to improve continence to a satisfactory level.

The SNS therapy has traditionally been applied as a two step procedure. Firstly, a 3-4 week test-period, often with a permanent electrode with tines, followed by permanent implantation if at least a 50% symptom reduction has been obtained during the test stimulation.

In a selected patient group(idiopathic faecal incontinence or incontinence as a result of an external anal sphincter tear (<160 degrees)) we have evidence that 90% of patients will have a successful test period (≥50% reduction in incontinence episodes). If preoperative there is motor response on at least 3 out of 4 poles on the lead, at a threshold ≤1.5 mAMP(unpublished data, submitted for publication) .

Thus, only 10% of the patients have the lead explanted after 3 to 4 weeks. In 90% of the patients a pacemaker is implanted after the test period, these patients will have an additional operation that could have been avoided if they had the permanent pacemaker implanted at the first stage.

Hypotheses In a selected patient group suffering from faecal incontinence a one-stage permanent implant will be possible. The functional results will be improved as more time can be spent finding the optimal pacemaker settings as the risk of infection is reduced compared to the stage implant. One-Stage implantation gives the opportunity to test the amount of placebo effect with SNS.

During the first 3 months postoperative patients will be randomized to either stimulation amplitude set at 90% of sensory threshold (control group) or 3 periods of stimulation at 0.05v (placebo), 50% and 90% of sensory threshold. Patients are randomized. After the initial 3 months the stimulation amplitude is increased to sensory threshold. After six months the project ends and the number of patients achieving the 50% improvement in incontinence episodes are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Informed consent
* Idiopathic faecal incontinence or incontinence following external sphincter tear ≤ 160 degrees.
* ≥ one faecal incontinence episode after optimized conservative treatment.
* Ability to use the patient programmer.

Exclusion Criteria:

* Pregnancy
* Diabetes
* Neurological diseases, including spinal cord injuries
* Pelvic irradiation
* Rectal resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Bowel Habit Diary changes | 12 weeks
  Change in number of incontinence episodes(Bowel Habit diary - ≥50% reduction in fecal incontinence episodes), compared to baseline.
Bowel Habit Diary changes | 4 weeks
  Change in number of incontinence episodes(Bowel Habit diary - ≥50% reduction in fecal incontinence episodes), compared to baseline.

SECONDARY OUTCOMES:
Bowel Habit Diary | 24 weeks
  Change in number of incontinence episodes(Bowel Habit diary - ≥50% reduction in fecal incontinence episodes), compared to baseline.
Functional outcome measure - Wexner Incontinence score | 4, 8, 12, and 24 weeks
  Changes in Wexner incontinence score, compared to baseline.
Functional outcome measure - St. Marks incontinence score | 4, 8, 12, and 24 weeks
  Changes in St. Marks incontinence score, compared to baseline.
Quality of Life FI - specific | 4, 8, 12, and 24 weeks
  Changes in Rockwood Faecal Incontinence Quality of Life score, compared to baseline
Changes in functional outcome - Urin incontinence (UI). | 4, 8, 12, and 24 weeks
  ICIQ_UI Short form,
Visual analogue score (VAS score): patients overall satisfaction | 4, 8, 12, and 24 weeks
  VAS-score (0-100) for patients satisfaction with overall:
  * Social function
  * Bowel function
  * Quality of life Baseline value used as reference
Anal physiology test | baseline, 4,8,12 and 25 weeks after implantation(Only in patients implanted in Aarhus, Denmark)
  Functional Lumen Imaging Probe (endoFLIP) and anal sensibility. The endoFLIP allows dynamic examination of the geometry and segmental distensibility properties of the anal canal by simultaneous measurement of anal pressure(PSI) and luminal cross sectional areas (CSAs) at 16 points along the length of the anal canal

CONTACTS AND LOCATIONS:
Overall Officials: Jakob K. Jakobsen, MD. Ph.D., Principal Investigator — Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital
Locations (1):
- Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All participants in the study group have access to the data and if agreed in the study group sub-analysis can be made after the trial has ended.